CLINICAL TRIAL: NCT02929537
Title: Transformation and Application of Diagnosis and Treatment Programs for COPD Based on Chronic Obstructive Pulmonary Disease Registration Research in China
Brief Title: China Chronic Obstructive Pulmonary Disease Registration Research
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Henan University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: COPD registration
Record Dates: First submitted 2015-09-29; First posted 2016-10-11 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Pulmonary Disease, Chronic Obstructive; registration research; Medicine, Chinese Traditional
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Western medicine: Patients in this group only choose conventional medicine treatment based on the classes of medications recommended by 2015 GOLD for COPD.
- Traditional Chinese Medicine: Patients in this group only choose conventional medicine treatment based on the Chinese Treatment Guidelines for COPD.
- Integrative Medicine: Patients in this group choose western medicine and Traditional Chinese Medicine.

SUMMARY:
With the comparative effectiveness research methods and hospital registration study approach, the purpose of this study is to objectively record the methods, efficacy and its influencing factors of COPD commonly used treatment methods/programs (Western medicine, Traditional Chinese Medicine and Integrative Medicine) in the actual medical environment, analysis of application characteristics for the different programs, and provide the basis for its revision and promotion. It is a first registration study for COPD in China.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a major disease of harm public health seriously. Although different treatment methods / programs (Western medicine, Traditional Chinese Medicine and Integrative Medicine) exist and are being developed to relieve symptoms and reduce mortality in COPD, most have only been studied in randomized controlled trials (RCT).

Most RCT study patients usually require a single disease, the use of standard treatment and a single intervention to evaluate interventions in an ideal state can achieve maximum effect,that is theoretical effect, it is difficult to provide the evidence of practical clinical efficacy or effectiveness. Secondly, RCT often require strict inclusion and exclusion criteria, resulting in inadequate representation of the study, thus limiting its conclusions spread to overall. There are some challenges for different treatment methods on the actual effect of the patients in the evaluation of conventional medical practice with RCT.

Real World Research based on clinical practice pay close attention highly in response to these problems, and the registry study had been applied widely in clinical practice. With the comparative effectiveness research methods and hospital registration study approach, based on the classes of medications recommended by 2014 GOLD and Chinese Treatment Guidelines for COPD, the purpose of this study is to objectively record the methods, efficacy and its influencing factors of COPD commonly used treatment methods/programs (Western medicine, Traditional Chinese Medicine and Integrative Medicine) in the actual medical environment, analysis of application characteristics for the different programs, and provide the basis for its revision and promotion. This is a first registration study for COPD in China.

ELIGIBILITY:
Inclusion Criteria:

* A confirmed diagnosis of COPD.
* With the informed consent signed.

Exclusion Criteria:

* Pregnant or breast-feeding women.
* Any psychiatric condition rendering the patient unable to understand the nature, scope and possible consequences of the study .
* Malignancy for which patient has undergone resection, radiation therapy or chemotherapy within the last 5 years.
* Complicated with respiratory disorders other than COPD (e.g., lung fibrosis, pulmonary thromboembolic).
* Complicated with heart failure (NYHA Class III or IV),or myocardial infarction within six months.
* Complicated with serious hepatic and renal diseases (liver cirrhosis, portal hypertension, bleeding of varicose veins, dialysis, or renal transplantation).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Peoples are diagnosed with Chronic Obstructive Pulmonary Disease (COPD).
Sampling Method: Non-Probability Sample
Enrollment: 3012 (Estimated)
Dates: Start 2015-05; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
The frequency of exacerbation | Change from Baseline in the frequency of exacerbation at the months 3, 6, 9, 12, 15, 18, 21 and 24.

SECONDARY OUTCOMES:
all cause mortality | through study completion, an average of 1 year
Forced expiratory volume in one second,FEV1 | Change from Baseline in the FEV1 at the months 6, 12, 18 and 24.
Dyspnea | Change from Baseline in the mMRC at the months 3, 6, 9, 12, 15, 18, 21 and 24.
  Using modified british medical research council (mMRC) to assess the degree of dyspnea in patients with COPD, and how this changes over time.
Symptoms | Change from Baseline in the CAT at the months 6, 12, 18 and 24.
  Using the COPD Assessment Test (CAT) as a comprehensive measure of symptoms.
Quality of life | Change from Baseline in the SF-36 at the months 6, 12, 18 and 24.
  Using the Chinese version of the 36-item Short Form Health Survey (SF-36) to measure quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Jiansheng Li, doctor, Study Chair — The First Affiliated Hospital of Henan University of Traditional Chinese Medicine